CLINICAL TRIAL: NCT07278011
Title: The Investigation of TAAR1 and JAK/STAT Pathway Gene Expression and Protein Levels in Inflamed Skin Tissue Samples From Patients With Hidradenitis Suppurativa
Brief Title: Molecular Evaluation of TAAR1 and JAK/STAT Pathway in Hidradenitis Suppurativa
Status: Completed | Type: Observational
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Gülden Karakalem, MD, Dermatology Resident, Trakya University
Other Study IDs: 2025/47; TÜTF-GOBAEK 2024/367 (Other: Trakya University Scientific Research Projects Unit)
Record Dates: First submitted 2025-11-30; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Hidradenitis Suppurativa (HS); Skin Inflammation
Keywords: Hidradenitis Suppurativa; TAAR1; JAK; STAT; SOCS; İnflammation
MeSH Terms: conditions — Hidradenitis Suppurativa; Dermatitis; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HS lesional skin group: Lesional skin biopsy samples were obtained from patients diagnosed with hidradenitis suppurativa. All samples were collected as part of routine clinical evaluation. No treatment interventions were performed as part of the study protocol.
- HS perilesional skin group: Perilesional (non-lesional) skin biopsy samples were obtained from patients diagnosed with hidradenitis suppurativa. Samples were collected from areas adjacent to active lesions during routine clinical evaluation. No procedures were performed as part of the study protocol.
- Healty control skin group: Skin biopsy samples were obtained from healthy individuals without inflammatory skin disease as a control group. The samples were collected solely for comparative molecular analysis. No intervention for treatment was performed.

SUMMARY:
This observational translational study aims to investigate gene and protein expression in lesional and perilesional skin of patients with Hidradenitis Suppurativa (HS) compared to controls. Skin biopsies were collected from 15 HS patients and 15 age- and sex-matched healthy controls. Gene expression of 15 selected proteins was analyzed using qRT-PCR, while protein levels of 4 targets were assessed by Western blot. The study seeks to identify molecular pathways involved in HS pathogenesis and potential biomarkers for disease severity.

DETAILED DESCRIPTION:
Hidradenitis suppurativa (HS) is a chronic, recurrent, inflammatory skin disease affecting areas rich in apocrine glands, characterized by painful nodules, abscesses, sinus tracts, and scar formation. Current evidence indicates that dysregulation of immune signaling pathways plays a central role in the pathogenesis of HS. Among these pathways, the JAK/STAT signaling cascade plays a role in the increase of the inflammatory response, while Trace Amine-Associated Receptor 1 (TAAR1), a G protein-coupled receptor, has recently been found to be associated with immune modulation. However, to our knowledge, the role of TAAR1 in HS has not been investigated before.

This observational study aimed to investigate the expression of genes and protein levels associated with the TAAR1 and JAK/STAT signaling pathways in patients with hidradenitis suppurativa. Lesional and perilesional skin biopsies were obtained from patients diagnosed with HS, and skin biopsy samples were obtained from healthy control individuals without inflammatory skin disease. Molecular analyses were performed to evaluate gene expression and protein levels.

The primary objective of the study was to compare the expression patterns of markers associated with the TAAR1 and JAK/STAT pathways between HS lesion skin, perilesion skin, and healthy control skin.

All participants were monitored in accordance with routine clinical practice, and no therapeutic intervention was applied within the scope of the study protocol. The study was conducted in accordance with the principles of the Helsinki Declaration, approved by the local Clinical Research Ethics Committee, and written informed consent was obtained from all participants prior to their inclusion in the study.

It is expected that the findings from this study will contribute to a better understanding of the molecular mechanisms of hidradenitis suppurativa and provide a scientific basis for targeted treatment approaches in the future.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years. Ability to read and write. For the patient group: clinical and/or histopathological diagnosis of hidradenitis suppurativa for at least 6 months.

No use of topical treatments within the last 2 weeks, conventional systemic treatments within the last 1 month, or biologic therapies within the last 3 months prior to enrollment.

Not pregnant at the time of enrollment. Absence of known immunosuppression or malignancy.

For the control group: healthy individuals aged ≥18 years without any autoimmune or inflammatory disease, matched to the hidradenitis suppurativa group in terms of age, sex, and metabolic characteristics, who presented for benign nevus excision at the Trakya University Medical Faculty Department of Dermatology.

Exclusion Criteria:

* Presence of any autoimmune or inflammatory disease other than hidradenitis suppurativa.

Current pregnancy. Known immunosuppression. History of malignancy. Use of topical, systemic conventional, or biologic treatments outside the defined washout periods.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 years and older with a clinical and/or histopathological diagnosis of hidradenitis suppurativa, as well as healthy control individuals aged 18 years and older without autoimmune or inflammatory disease. Healthy controls were selected to be similar to the hidradenitis suppurativa group in terms of age, sex, and metabolic characteristics. Control participants were recruited among individuals presenting for benign nevus excision at the Trakya University Medical Faculty Department of Dermatology.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2025-11-21 (Actual)

PRIMARY OUTCOMES:
Expression levels of TAAR1 and JAK/STAT pathway markers in skin tissue | At the time of molecular analysis (September 2025)
  To evaluate and compare the gene and protein expression levels of TAAR1 and selected JAK/STAT pathway components in lesion and perilesion skin samples from patients diagnosed with hidradenitis suppurativa and in healthy control skin samples using molecular methods.

CONTACTS AND LOCATIONS:
Overall Officials: Yıldız Gürsel Ürün, MD, Study Chair — Trakya University; Zeynep Banu Doğanlar, PhD, Study Director — Trakya University
Locations (1):
- Trakya University Medical Faculty, Department of Dermatology, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy and confidentiality considerations and in accordance with the approved ethics committee protocol.